CLINICAL TRIAL: NCT01456572
Title: Gastric and Intestinal Satiation in Obese and Normal Weight Healthy People
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: EKBB 122/09
Record Dates: First submitted 2011-09-29; First posted 2011-10-20 (Estimated); Last update posted 2011-10-20 (Estimated); Status verified 2011-10

CONDITIONS: Endocrine System Diseases
Keywords: glucagon-like peptide-1; peptide tyrosine tyrosine; ghrelin; stomach; small intestine; gastric emptying
MeSH Terms: conditions — Endocrine System Diseases | interventions — Ensure Plus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- satiation_obese weight (Active Comparator): Obese subjects will receive a complex nutrient drink (Ensure Plus; 17 % protein, 30 % fat and 53 % carbohydrate, 1 kcal/mL). Nutrient intake will be stopped when subjects had reached maximal or unbearable satiation; the time needed to reach the maximal level of satiation (tmax) and the quantity of volume drunk will be recorded and calorie intake calculated.
  Interventions: Dietary Supplement: ensure plus
- gastric emptying_obese weight (Active Comparator): Obese subjects will receive a standardized meal, consisting of two scrambled eggs (cooked with 10 g butter), placed on two slices of whole wheat bread and 200 mL of milk (in total: 468 kcal). The test meal will be labeled with 100 mg of 13C-octanoic acid for determination of gastric emptying.
  Interventions: Dietary Supplement: standardized test meal
- gastric emptying_normal weight (Placebo Comparator): Normal weight subjects will receive a standardized meal, consisting of two scrambled eggs (cooked with 10 g butter), placed on two slices of whole wheat bread and 200 mL of milk (in total: 468 kcal). The test meal will be labeled with 100 mg of 13C-octanoic acid for determination of gastric emptying.
  Interventions: Dietary Supplement: standardized test meal
- satiation_normal weight (Placebo Comparator): Normal weight subjects will receive a complex nutrient drink (Ensure Plus; 17 % protein, 30 % fat and 53 % carbohydrate, 1 kcal/mL). Nutrient intake will be stopped when subjects had reached maximal or unbearable satiation; the time needed to reach the maximal level of satiation (tmax) and the quantity of volume drunk will be recorded and calorie intake calculated.
  Interventions: Dietary Supplement: ensure plus
- hormone profiles_obese weight (Active Comparator): Obese subjects will receive 500 mL of a complex nutrient drink (Ensure Plus; 17 % protein, 30 % fat and 53 % carbohydrate). At regular time intervals fasting and post-prandial blood samples will be collected.
  Interventions: Dietary Supplement: ensure plus
- hormone profiles_normal weight (Placebo Comparator): Normal weight subjects will receive 500 mL of a complex nutrient drink (Ensure Plus; 17 % protein, 30 % fat and 53 % carbohydrate). At regular time intervals fasting and post-prandial blood samples will be collected.
  Interventions: Dietary Supplement: ensure plus

INTERVENTIONS:
Dietary Supplement: ensure plus — 17 % protein, 30 % fat and 53 % carbohydrate; 1 kcal/mL
  Arms: hormone profiles_normal weight; hormone profiles_obese weight; satiation_normal weight; satiation_obese weight
Dietary Supplement: standardized test meal — scrambled eggs, two slices of whole wheat bread, 200 mL of milk and labeled with 13C-octanoic acid
  Arms: gastric emptying_normal weight; gastric emptying_obese weight

SUMMARY:
The purpose of this study is to determine the reciprocal control between gastric functions and intestinal parameters in the development of satiation in obese people.

DETAILED DESCRIPTION:
Obesity has reached pandemic proportions, obesity-associated complications are extensive and the current treatment options are limited. These facts demonstrate the need for an improved understanding of the pathogenesis of obesity. The gastrointestinal tract plays a key element in the control of satiation; discrepancies exist, however, for the role of gastric and intestinal parameters in the control of satiation in relation to body mass. To achieve a comprehensive understanding for the reciprocal control between gastric functions and intestinal parameters in the development of satiation in obese people the investigators will compare satiation parameters, gastric emptying and plasma glucagon-like peptide-1 (GLP-1), peptide tyrosine tyrosine (PYY) and ghrelin levels between normal and obese healthy volunteers.

Time needed to reach the level of satiation and total calorie intake will be measured by a standardized nutrient drink test; gastric emptying of solids by a 13C-octanoic acid breath test; and plasma GLP-1, PYY and ghrelin levels will be measured after a standardized nutrient drink.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects
* age 18-45

Exclusion Criteria:

* smoking
* substance abuse
* regular intake of medication
* medical or psychiatric illness
* gastrointestinal disorders or food allergies

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2007-01; Primary Completion 2011-02 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
gastrointestinal peptide secretion | 2 hours blood sampling

SECONDARY OUTCOMES:
gastric emptying | 240 minutes end-expiratory breath sample collection
time needed to reach the level of satiation | up to 30 min
total calorie intake | up to 30 min

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Beglinger, MD, Principal Investigator — Phase 1 Research Unit, University Hospital Basel
Locations (1):
- University Hospital Basel, Phase 1 Research Unit, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Derived] Meyer-Gerspach AC, Wolnerhanssen B, Beglinger B, Nessenius F, Napitupulu M, Schulte FH, Steinert RE, Beglinger C. Gastric and intestinal satiation in obese and normal weight healthy people. Physiol Behav. 2014 Apr 22;129:265-71. doi: 10.1016/j.physbeh.2014.02.043. Epub 2014 Feb 28. PMID 24582673